CLINICAL TRIAL: NCT02697747
Title: Identification of L3-L4 Interspace in Parturients
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Phillip Hess, Staff Anesthesiologist, Beth Israel Deaconess Medical Center
Other Study IDs: 2015P000225
Record Dates: First submitted 2015-11-16; First posted 2016-03-03 (Estimated); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Healthy
Keywords: Ultrasound; Palpation; Analgesia; Epidural
MeSH Terms: conditions — Agnosia | interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ultrasound education: Training in the use of ultrasound to identify the L3-L4 interspace
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — Educational intervention in the use of ultrasound to identify landmarks

SUMMARY:
The investigators hypothesize that teaching ultrasound sonoanatomy to identify the L3-L4 interspace will improve resident's long term skill to correctly identify the interspace as compared to palpation alone.

DETAILED DESCRIPTION:
This will be an observational education based study to improve anesthesiology resident's ability to correctly identify the L3-L4 interspace. Residents who agree to participate in the study will be trained using ultrasound to identify the L3-L4 interspace during their rotation on the obstetric anesthesia service. Training will include using the ultrasound to correlate the surface palpation with the underlying structures. This will be supplemented with teaching videos and literature. The training will be performed for the first three weeks of the four week rotation.

After undergoing this training program, during the fourth week of the rotation, the residents will be asked to perform palpation identification of the L3-L4 interspace on parturients. Ultrasound will be used to assess the accuracy of the identified level. These assessments will repeated at six and 12 months to assess whether the skill has been retained.

ELIGIBILITY:
Inclusion Criteria:

* term gestation (at least 38 weeks gestation)

Exclusion Criteria:

* Prior back surgery
* Previously diagnosed skeletal deformities such as scoliosis
* BMI greater than 40
* Height less than 60 inches
* Patient discomfort requiring immediate analgesia

Ages: 12 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant female patients.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2015-11; Primary Completion 2020-12 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Accuracy measured as percentage of cases where the L3-4 vertebral interspace is identified correctly | 1 month
  Percentage of cases where the L3-4 vertebral interspace is identified correctly

SECONDARY OUTCOMES:
Durability measured as percentage of cases where the L3-4 vertebral interspace is identified correctly | 6 months and 12 months
  percentage of cases where the L3-4 interspace is identified correctly at 6 months and again at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Philip E Hess, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No